CLINICAL TRIAL: NCT02327936
Title: Efficacy and Tolerability of Fesoterodine and Oxybutynin XL for Overactive Bladder Syndrome in Children: a Comparative Study.
Brief Title: Fesoterodine and Oxybutynin XL for Overactive Bladder Syndrome in Children
Acronym: FOXY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stéphane Bolduc (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Stéphane Bolduc, MD, FRCSC, CHU de Quebec-Universite Laval
Organization: CHU de Quebec-Universite Laval (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FOXY2014
Record Dates: First submitted 2014-12-10; First posted 2014-12-31 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fesoterodine 4mg (Experimental): Fesoterodine 4 mg Po Die, dose could be increased to 8mg Po Die after 4 weeks, for a total of 8 weeks
  Interventions: Drug: Fesoterodine
- Oxybutynin XL 10mg (Active Comparator): Oxybutynin XL 10 mg Po Die, dose could be increased to 20 mg Po Die after 4 weeks, for a total of 8 weeks
  Interventions: Drug: Oxybutynin XL

INTERVENTIONS:
Drug: Fesoterodine — Administer medication to patients with overactive bladder
  Other Names: Toviaz
  Arms: Fesoterodine 4mg
Drug: Oxybutynin XL — Administer medication to patients with overactive bladder
  Other Names: Ditropan XL
  Arms: Oxybutynin XL 10mg

SUMMARY:
The purpose of this study is to evaluate the tolerability of Fesoterodine and Oxytbutynin XL and to compare their efficacy for overactive bladder syndrome in children.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a highly prevalent disorder in the pediatric population. This condition comprises many urinary symptoms, such as urgency, increased daytime frequency of micturition, urge incontinence and nocturia1, 2. These symptoms are especially troublesome for the pediatric patients and their family since it causes embarrassment and it limits everyday activities and impairs children's development. Furthermore, serious complications are seen if this condition is not treated properly, as urinary tract infection, vesico-ureteral reflux and dysfunctional voiding. Antimuscarinic agents are the current pharmacologic mainstay for OAB. Many side effects are reported with the clinical use of antimuscarinics. In the last years, Fesoterodine, a new antimuscarinic, has been developed for the treatment of OAB. Studies show significant improvement of clinical symptoms in adults with OAB and fewer side effects. The outcomes for the pediatric population remain unknown due to lack of studies. Antimuscarinic agents are the mainstay of the current treatment of OAB. Oxybutynin is the most widely antimuscarinic agent used in the pediatric population and is the only molecule approved by Health Canada for children with OAB. However, some patients have a suboptimal response to antimuscarinic and many experience side effects. Children with OAB therefore represent a disease population with a need for an alternative effective, safe and well-tolerated therapy to help manage the overactive detrusor, reducing or preventing incontinence. Fesoterodine is a new antimuscarinic drug available as a prolonged release (PR) tablet formulation, and is approved in Europe, Canada and the USA at doses of 4 mg and 8 mg once daily for the treatment of OAB in adults; it is not approved for use in the pediatric population. Before randomization, subjects will undergo 2 weeks of urotherapy. At the end of these 2 weeks, the inclusion and exclusion criteria will be reassessed and the subjects admissible for the study will be randomized for a 8 week-treatment period during which the urotherapy will be continued. Eligible subjects will be randomized to 8 weeks of single-blind treatment with Fesoterodine 4 mg Po Die or Oxybutynin XL 10 mg Po Die. At the end of the 8 week-treatment period, subjects will stop their current therapy for one week. At week 9, both cohorts will do a cross over. The cohort on Fesoterodine will be on Oxybutynin XL and vice versa. After 4 weeks on any given medication, the possibility of up-titration will be assessed. On a telephone interview with the research nurse, patients and parents will be questioned on compliance, tolerability and efficacy. If the patient is taking the medication ≥80% of the time, does not have any significant side effects and still has significant OAB symptoms, the investigators will offer a dose increase (Fesoterodine 8mg or Oxybutynin XL 20mg daily). If accepted, the medication will be provided with instructions to report any new side effects. Oxybutynin XL (Ditropan XL) is the extended release and once a day formulation of Oxybutynin (actual gold standard for OAB in children). By using this formulation with children who can swallow pills, the control group has the same once a day regimen as Fesoterodine (Toviaz), thus avoiding this possible bias. The bid or tid immediate release formulation is known to create more side effects and decreases the compliance (sometime hard to administer the afternoon dose to children at school).

Subjects will complete a 3-day voiding diary prior to each medical visit to assess the efficacy of the single-blind treatment and urotherapy. Visits will be done on week -2, 0, 8 and 17 (+/- 5 days)

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 5 years old and ≤14 years old
* OAB diagnostic according to the International Children Continence Society (ICCS) and less than 65% of the expected mean bladder capacity for age is confirmed (30 + (age in years x 30) mL) on a 3-day voiding diary.
* Weight and height are within the normal percentile (3rd to 97th percentile) and weight is ≥ 20 kg (3rd percentile of a 8 y.o. child, boy or girl), according to the CDC growth chart
* Ability to swallow pills
* Subjects/parents (vs. legal guardian) agree to participate to the following study and sign the informed consent
* Subjects/parents (vs. legal guardian) are able to comply with the study requirements and with the medication restrictions.

Female subjects of childbearing potential must have a negative serum or urine pregnancy test at enrollment and must agree to maintain highly effective birth control during the study. Sexually active male subjects agree to use a barrier method of birth control with female partner for the duration of the study and at least one month after ending study treatment. Sexually active male subjects agree to use a condom for the duration of the study and for at least one month after ending study treatment and the female partner to use a reliable form of birth control for the duration of the study and for at least one month after ending study treatment.

Exclusion Criteria:

* Subject has a diagnostic of dysfunctional voiding
* Post-voiding residue > 20 cc
* Polyuria (> 75 ml/kg/b.w./24 hours)
* Nephrogenic of central diabetes insipidus
* Constipation at screening (if the patient is treated and the treatment is successful, the patient will be eligible to the study)
* Urinary tract infection at visit 2-3-4. If UTI is present at the screening visit, the UTI must be treated and the success of the treatment must be documented with a negative urinalysis at visit 2.
* QTc interval greater than 460 ms, or any increase of 30 ms on follow-up EKG (mean of 6 separate EKG-3 from visit week-2 and 3 from visit week 0). If a patient meets those criteria in the first month (initial dose), he will be excluded from the study. If the QTc change is noted after the up-titration, the dose will be decreased and EKG will be repeated within 1 week to ensure normalization of QTc.
* Clinically significant unstable medical condition or disorder
* Subject is pregnant or intends to become pregnant
* Serum creatinin more than or equal to 2 times the upper limit of normal
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than or equal to 2 times ULN, or bilirubin more than or equal to 1.5 times ULN.
* Known hypersensitivity to Oxybutynin or Fesoterodine or any contraindication to the use of those 2 molecules, in accordance to the product monography (to the exception of pediatric age).
* Subject is taking medication that interact with Fesoterodine and this medication can't be discontinued (see appendix 1 of excluded drugs)
* Known urological pathology other than OAB that could explain urinary symptoms (as bladder stone…)
* Non-treated or non-controlled arterial hypertension

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2014-12; Primary Completion 2018-03 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of Fesoterodine and Oxybutynin XL | 4 months
  Side effects: the number of patients in each arm presenting side effects of grade 1, 2 and 3 (mild, moderate, severe).
  Between study arms, for cardiovascular safety: mean difference in blood pressure, mean difference in heart rate, mean difference in QTcB.
  * Vital signs (blood pressure and heart rate),
    * Increase of more than 20% of heart rate at rest
    * Variation in blood pressure: systolic ±20 mmHg, diastolic ±15 mmHg
  * Or symptoms suggesting it, without reaching those variations. o Parameters to be measure at each visit but particularly at visit 2 (Week 0, first dose on site), to be obtained before and 1 hour after taking the medication.
  Blood tests profile comparing number of subjects with significant changes: Blood work (including hepatic and renal workups, electrolytes, Hb-Ht).

SECONDARY OUTCOMES:
Number of Participants with Improved Overactive Bladder Symptoms as a Measure of Efficacy of Fesoterodine and Oxybutynin XL | 4 months
  Improved symptoms: Change from baseline to final voiding diary (after completion of each treatment on week 8 and week 17) in mean volume per micturition (first micturition of the day excluded).
Number of urgency and urinary incontinence episodes as a Measure of Efficacy of Fesoterodine and Oxybutynin XL | 4 months
  * Mean number of daytime incontinence per 24 h.
  * Mean number of nighttime incontinence per 24 h.
  * Mean number of grade 2 and 3 urgency episodes (according to the CUA voiding diary; 0-3) per 24 h.
  * Mean number of micturition per 24 h.
  * Effectiveness will also be assessed using the Patient Perception of Bladder Condition (PPBC) scale on a 6-point scale ranging from 1 to 6, at study initiation and every visit.
  * Results will be documented based on subjective relief of symptoms and objective voiding diaries following the ICCS classification.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Bolduc, MD, Principal Investigator — CHU de Québec-Université Laval

IPD SHARING:
Plan to Share IPD: Yes
Publication to be submitted in peer reviewed journal, end of 2019
Supporting Information: CSR
Time Frame: after publication
Access Criteria: online via journal